CLINICAL TRIAL: NCT01038960
Title: Exercise Training to Reduce Ventricular Arrhythmia in Heart Failure Patients With ICD - The Ethic Study
Brief Title: Exercise Training in ICD Recipients; Effect on Therapy Delivered, Depression and Anxiety
Acronym: ETHIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Stavanger Health Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETHIC-SUS-AIL-09; 068.08 (Registry Identifier: Norwegian Social Science Data Services)
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Ventricular Tachycardia
Keywords: ICD, training
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise training (Experimental): training
  Interventions: Behavioral: Exercise training
- Not training (No Intervention): No organized training

INTERVENTIONS:
Behavioral: Exercise training — 3 months supervised interval training
  Other Names: ICD, exercise training
  Arms: Exercise training

SUMMARY:
Interventional study in patients with ICD. Controlled, open intervention with exercise training. Assessment of changes in physiological and psychological parameters.

DETAILED DESCRIPTION:
ICD therapy with DC shock is associated with impaired quality of life and development of anxiety and depression. In a selected group of patients with ICD the intervention with organized high intensity training is evaluated. Peak VO2, inflammatory profile, performed interventions by the ICD and psychological profile is assessed. In addition a qualitative evaluation using interviews is performed.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: Age 18 years or above, documented coronary heart disease, myocardial scar tissue verified by CMR, implanted ICD

Exclusion Criteria:

* Planned revascularisation by bypass surgery or percutaneous coronary intervention following the ICD implantation, planned arrhythmia ablation, long QT-syndrome, Brugada syndrome, WPW syndrome, Drug-induced torsades, catecholaminergic polymorphic ventricular tachycardia, Hypertrophic cardiomyopathy right ventricular cardiomyopathy, dilated cardiomyopathy, Aortic stenosis, mitral valve prolapse, anomalous origin of coronary arteries, Myocardial bridging, ongoing myocarditis, recent chest trauma,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Therapy delivered from ICD, Anxiety score, functional status | 3 months

SECONDARY OUTCOMES:
HRV, Endothelial function | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alf Inge Larsen, MD, PhD, Principal Investigator — University of Bergen
Locations (1):
- Stavanger Health Research, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: No